CLINICAL TRIAL: NCT02125136
Title: Prospective Randomized Multicenter Phase II Trial to Investigate Intensified Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Cancer
Brief Title: Trial to Investigate Intensified Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Cancer
Acronym: NEOLAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Celgene Corporation (Industry); ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-PAK-0113; AX-CL-PANC-PI-003324 (Other Grant/Funding Number: Celgene); 2013-004796-12 (EudraCT Number)
Record Dates: First submitted 2014-04-11; First posted 2014-04-29 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Ductal Adenocarcinoma of the Pancreas
Keywords: unresectable; borderline resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gem/nab-Pac (Experimental): 2 further cycles Gem/nab-Pac (duration of each cycle 28 days)
  Interventions: Drug: Gem/nab-Pac
- FOLFIFINOX (Experimental): 4 cycles combination therapy with 5-fluorouracil/folinic acid, irinotecan, oxaliplatin (FOLFIFINOX) - duration of each cycle 14 days
  Interventions: Drug: FOLFIFINOX

INTERVENTIONS:
Drug: Gem/nab-Pac — All patient receive:
  2 cycles gemcitabine/nab-paclitaxel ([Gem/nab-Pac]; duration of each cycle 28 days)
  Then:
  Nab-paclitaxel 125 mg/m2, IV infusion over 30 minutes, followed by gemcitabine 1000 mg/m2 as a 30-minute IV infusion on D1, D8, D15 of each 28-day cycle
  Arms: Gem/nab-Pac
Drug: FOLFIFINOX — All patient receive:
  2 cycles gemcitabine/nab-paclitaxel ([Gem/nab-Pac]; duration of each cycle 28 days)
  Then:
  Oxaliplatin 85 mg/m2, given as a 2-hour intravenous infusion D1 Folinic acid 400 mg/m2, given as a 2-hour intravenous infusion D1 Irinotecan 180 mg/m2, given as a 90-minutes intravenous infusion D1 (application through a Y-connector parallel to infusion of folinic acid or 30 minutes after start of folinic acid possible) Fluorouracil 400 mg/m2, administered by intravenous bolus, followed by a continuous intravenous infusion of fluorouracil 2400 mg/m2 over a 46-hour period D1.
  To be repeated on D1 of each cycle.
  Arms: FOLFIFINOX

SUMMARY:
The aim ot the study is to investigate the efficacy and safety of two new intensified chemotherapy regimens (gemcitabine (Gem)/nab- paclitaxel (PAC), FOLFIRINOX) as neoadjuvant chemotherapy protocol in locally advanced, non-metastatic pancreatic cancer (LAPC) and consecutive conversion of the tumor to resectability.

DETAILED DESCRIPTION:
This is a prospective open randomized multicenter phase II trial with two arms.

Patients suffering from histologically confirmed LAPC (and assessed as unresectable or borderline resectable according to National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines "pancreatic adenocarcinoma" version 1.2013) without metastases will receive two different neoadjuvant treatment regimens:

First all patients receive two cycles Gem/nab-PAC (duration of each cycle 28 days) as neoadjuvant chemotherapy in equal measure and a first restaging is performed after these two cycles based on imaging criteria. If there is no progression according to Response evaluation criteria in solid tumors (RECIST 1.1) criteria at the first restaging, the patients are randomized in a 1:1 relation to:

Two further cycles Gem/nab-PAC (duration of each cycle 28 days). or Four further cycles FOLFIRINOX (duration of each cycle 14 days). After the neoadjuvant chemotherapy a 2nd restaging is performed based on imaging criteria. All patients without progression at this restaging or at an earlier time point undergo obligatory exploratory laparotomy irrespective of imaging criteria to assess resectability. If they are evaluated as converted to resectable during this exploratory laparotomy, pancreas resection in curative intent will be performed. All patients with successful R0 or R1 pancreatic resection will receive three further cycles adjuvant chemotherapy with Gem/nab-PAC. Adjuvant chemotherapy will start within 4 to 8 weeks after pancreatic resection surgery.

Further treatment of patients with PD after 1st or 2nd restaging as well as patients with unresectable status based on exploratory laparotomy is under the discretion of the local investigators (e.g. second-line chemotherapy in case of distant relapse or local radiochemotherapy in case of local progression or definitive irresectability).

All patients are followed up for local recurrence, progression and survival until death or for at least one year after last application of study drugs whichever is sooner.

The translational research conducts exploratory analyses for potential biomarkers of possible prognostic or predictive value for efficacy of neoadjuvant chemotherapy in LAPC; including analyses of circulating tumor cells, molecular pathways of pancreatic adenocarcinoma including SPARC expression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years and ≤ 75 years of age
* Histologic or cytologic proven ductal adenocarcinoma of the pancreas (histologic confirmation of diagnosis is preferred)
* No distant metastases
* De novo, treatment-naïve unresectable or borderline resectable LAPC; evaluation of unresectable and borderline resectable status according to NCCN- Clinical Practice Guidelines in Oncology "pancreatic adenocarcinoma" version 1.2013. Applicable criterion/criteria have to be indicated.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Total bilirubin ≤ 2 mg/dL. Patients with a biliary stent may be included provided that bilirubin level after stent insertion decreased to ≤ 2 mg/dL and there is no cholangitis.
* Adequate renal, hepatic and bone marrow function, defined as
* Serum creatinine ≤ 1.25 x Upper limit of normal (ULN)
* Calculated creatinine clearance ≥ 60 mL/min according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Aspartate aminotransferase (AST)/(serum glutamic oxaloacetic transaminase)GOT and/or Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (GPT) ≤ 2.5 x ULN
* Partial thromboplastin time (PTT) ≤ 1.5 x ULN and Quick value ≥ 70%
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Haemoglobin ≥ 8g/dL
* Platelets ≥ 100 x 109/L
* Females of childbearing potential (FCBP) must have a negative pregnancy test within 7 days of the first application of study treatment and must agree to use effective contraceptive birth control measures (Pearl Index < 1) during the course of the trial and for at least 1 month after last application of study treatment.

A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 year, or unless she is surgically sterile.

* Males must agree not to father a child during the course of the trial and for at least 6 months after last administration of study drugs.
* Signed and dated informed consent before the start of any specific protocol procedures
* Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Evidence of distant metastases. In case of radiological suspicion of peritoneal carcinomatosis or ascites histological or cytological verification is required e.g. by means of exploratory laparoscopy
* Local relapse of the pancreatic adenocarcinoma prior treated with surgical resection
* Any previous treatment of the pancreatic carcinoma (radiotherapy, chemoradiotherapy, chemotherapy, targeted tumor therapy, local ablative therapy)
* Contraindication for pancreas resection (pancreatic head resection, distal pancreatectomy with splenectomy, or complete pancreatectomy)
* Larger surgical interventions within 4 weeks before study enrolment and/or diagnostic laparotomy with or without gastroenterostomy and with or without biliodigestive anastomosis within 2 weeks before first application of study treatment. Wound healing must be also completed before first application of study treatment.
* Known chronic diarrhoea
* Peripheral polyneuropathy > grade 1
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Medical history of interstitial lung disease (ILD) or pulmonary fibrosis
* Hypersensitivity against any of the study drugs (nab-paclitaxel, gemcitabine, oxaliplatin, irinotecan, 5-fluorouracil, folinic acid), or the ingredients of these drugs
* Active or uncontrolled bacterial, viral, or fungal infection that requires systemic treatment
* Known HIV- infection or active Hepatitis B virus (HBV)- or Hepatitis C virus (HCV) infection
* Convulsion disorder that requires anticonvulsive treatment
* Clinically significant cardiovascular or vascular disease or disorder ≤ 6 months before study enrolment (e.g. myocardial infarction, unstable angina pectoris, chronic heart failure New York Heart Association (NYHA) ≥ grade 2, uncontrolled arrhythmia, cerebral infarction)
* Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the study and his/her safety during the study or interfere with interpretation of study results e.g. severe hepatic, renal, pulmonary, metabolic, or psychiatric disorders
* Requirement for concomitant antiviral treatment with sorivudine or brivudine
* Requirement of immunosuppressive treatment
* Continuing anticoagulant therapy with coumarin derivatives (treatment with low-molecular weight heparin allowed)
* Continuing abuse of alcohol, drugs, or medical drugs
* Pregnant or breast feeding females
* Participation in any other clinical trial or treatment with any experimental drug within 28 days before enrolment to the study or during study participation until the end of treatment visit.
* Previous or concurrent malignant tumor disease other than underlying tumor disease with the exception of cervical cancer in situ, adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder tumors (Ta,Tis, and T1) or any curatively treated tumors > 5 years prior to enrolment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Conversion Rate | approx. 10 month
  To compare the effect of intensified neoadjuvant chemotherapy on conversion rate to resectability in LAPC.

SECONDARY OUTCOMES:
Safety | approx. 22 month
  evaluate safety and tolerability of intensified neoadjuvant chemotherapy
  * Exposure to study drugs
  * Type, incidence, and severity of adverse events
  * Dose reduction or discontinuation of study drugs due to adverse events
  * Laboratory parameters
objective tumour response rate | approx. 22 month
  assess objective tumour response rate (ORR) to intensified neoadjuvant chemotherapy Baseline tumor measurement(s) will be performed within 4 weeks before the first dose of study drug with either computed tomography (CT) including spiral CT or MRI according to investigator's choice and clinical practice at the respective trial site as done routinely also outside of clinical trial situations.The same method used at baseline must be used consistently for response assessment to neoadjuvant chemotherapy at the first restaging (after the first part of neoadjuvant chemotherapy) and the second restaging (after the second part of neoadjuvant chemotherapy) and thereafter.
disease control rate (DCR) | approx. 22 month
  assess disease control rate (DCR) after intensified neoadjuvant chemotherapy
CA 19-9 change | 10 month
  Assess carbohydrate antigen 19-9 (CA 19-9) change during/after neoadjuvant chemotherapy. In this trial, CA 19-9 change to neoadjuvant chemotherapy will be evaluated as decrease to the baseline level at the 1st and 2nd restaging.
R0 and R1 resections | 10 month
  assess rate of R0 and R1 resections
pathological responses | approx. 22 month
  assess rate of grade 3 + 4 pathological responses according to grading scheme of treatment responses by Evans in resected patients.
relapse-free survival (RFS) | approx. 22 month
  assess relapse-free survival (RFS): Relapse-free survival is the time from Day 1 after pancreatic resection to the date of relapse, defined as Day 1 after pancreatic resection to either local relapse of pancreatic cancer or occurrence of distant metastases. For each patient who is not known to have had a relapse as of the data-inclusion cut-off date for a particular analysis, time to relapse will be censored for that analysis at the date of the patient's last study visit prior to that cut-off date.
Progression-free survival (PFS) | approx. 2 years
  PFS is the time from Day 1 of the first cycle of neoadjuvant chemotherapy to date of objective disease progression or to death of any cause.
  For each patient who is not known to have had a progression as of the data-inclusion cut-off date for a particular analysis, time to progressive disease will be censored for that analysis at the date of the patient's last study visit prior to that cut-off date.
perioperative morbidity and mortality | 60 days
  assess perioperative morbidity and mortality
Tolerability | 10 month
  evaluate safety and tolerability of intensified neoadjuvant chemotherapy (see safety measure)
Overall Survival (OS) | approx. 22 month
  OS is the time from Day 1 of the first cycle of neoadjuvant chemotherapy to date of death from any cause.
  The rate of patients who have died from any cause after one year and two years, respectively will be assessed. For each patient for whom it is not known whether he died or is still alive until the data-inclusion cut-off date for a particular analysis, time to death of any cause will be censored for that analysis at the date of the patient's last study visit prior to that cut-off date.

CONTACTS AND LOCATIONS:
Overall Officials: Kunzmann Volker, Prof. Dr., Principal Investigator — Universitätsklinikum Würzburg/Comprehensive Cancer Center Mainfranken
Locations (1):
- Universitätsklinikum Würzburg/Comprehensive Cancer Center Mainfranken, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Hartlapp I, Valta-Seufzer D, Siveke JT, Algul H, Goekkurt E, Siegler G, Martens UM, Waldschmidt D, Pelzer U, Fuchs M, Kullmann F, Boeck S, Ettrich TJ, Held S, Keller R, Anger F, Germer CT, Stang A, Kimmel B, Heinemann V, Kunzmann V; German Pancreatic Cancer Group (AIO-PAK) and NEOLAP investigators. Prognostic and predictive value of CA 19-9 in locally advanced pancreatic cancer treated with multiagent induction chemotherapy: results from a prospective, multicenter phase II trial (NEOLAP-AIO-PAK-0113). ESMO Open. 2022 Aug;7(4):100552. doi: 10.1016/j.esmoop.2022.100552. Epub 2022 Aug 12. PMID 35970013
- [Derived] Kunzmann V, Siveke JT, Algul H, Goekkurt E, Siegler G, Martens U, Waldschmidt D, Pelzer U, Fuchs M, Kullmann F, Boeck S, Ettrich TJ, Held S, Keller R, Klein I, Germer CT, Stein H, Friess H, Bahra M, Jakobs R, Hartlapp I, Heinemann V; German Pancreatic Cancer Working Group (AIO-PAK) and NEOLAP investigators. Nab-paclitaxel plus gemcitabine versus nab-paclitaxel plus gemcitabine followed by FOLFIRINOX induction chemotherapy in locally advanced pancreatic cancer (NEOLAP-AIO-PAK-0113): a multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):128-138. doi: 10.1016/S2468-1253(20)30330-7. Epub 2020 Dec 16. PMID 33338442
- See also: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de